CLINICAL TRIAL: NCT06907290
Title: A Global, Randomized, Open-label, Multicenter, Phase 2b/3 Trial Evaluating BJT-778 vs Delayed Treatment for the Treatment of Chronic Hepatitis Delta Infection (AZURE-1)
Brief Title: A Trial Evaluating BJT-778 vs Delayed Treatment for the Treatment of Chronic Hepatitis Delta Infection
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Bluejay Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BJT-778-301
Record Dates: First submitted 2025-03-26; First posted 2025-04-02 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2026-01

CONDITIONS: Chronic Hepatitis D Infection
Keywords: Hepatitis Delta virus; HDV; Hepatitis D infection; Hepatitis D virus
MeSH Terms: conditions — Hepatitis D | interventions — Treatment Delay

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Brelovitug 300mg (Experimental): Dose - brelovitug 300 mg Frequency- once weekly
  Interventions: Drug: Brelovitug 300 mg
- Brelovitug 900mg (Experimental): Dose - brelovitug 900 mg Frequency- once every 4 weeks
  Interventions: Drug: Brelovitug 900 mg
- Delayed Treatment with brelovitug 300mg (Active Comparator): Dose - brelovitug 300 mg Frequency- 24 weeks of delayed treatment, then once weekly
  Interventions: Drug: Delayed Treatment with Brelovitug 300mg

INTERVENTIONS:
Drug: Brelovitug 300 mg — Route of administration- Subcutaneous Injection
  Arms: Brelovitug 300mg
Drug: Brelovitug 900 mg — Route of administration- Subcutaneous Injection
  Arms: Brelovitug 900mg
Drug: Delayed Treatment with Brelovitug 300mg — Route of administration- Subcutaneous Injection
  Arms: Delayed Treatment with brelovitug 300mg

SUMMARY:
This is a Phase 2b/3 study designed to evaluate the safety and efficacy of chronic treatment with brelovitug (a.k.a BJT-778; BTG) for chronic hepatitis delta virus (HDV) infection. The comparator in this study will be 24-weeks of delayed treatment. During the 24-weeks of delayed treatment, participants will complete the same visits and assessments as those randomized to initiate brelovitug immediately. At the completion of 24-week delayed treatment period, all participants will start treatment with brelovitug.

DETAILED DESCRIPTION:
Study will consist of 3 study arms. Approximately 150 participants will be randomized 2:2:1 to one of the following treatment arms:

* Arm 1: Participants randomized to Arm 1 will receive brelovitug 300 mg subcutaneously once weekly.
* Arm 2: Participants randomized to Arm 2 will receive brelovitug 900 mg subcutaneously once every 4 weeks.
* Arm 3: Participants randomized to Arm 3 will attend study clinic visits and delay treatment with brelovitug. At Week 24, all participants will receive brelovitug 300 mg subcutaneously once weekly.

ELIGIBILITY:
Inclusion Criteria:

* Willing and able to provide written informed consent.
* Chronic HDV infection
* HDV RNA >500 IU/mL at Screening.
* Abnormal ALT (>upper limit of normal) at Screening.
* Willing to take or already taking HBV nucleos(t)ide therapy

Exclusion Criteria:

* Pregnant or nursing females.
* Unwilling to comply with contraception requirements during the study.
* Difficulty with blood collection and/or poor venous access for the purposes of phlebotomy
* Presence of other liver disease(s) (does not include HBV or HDV infection) such as non-alcoholic steatohepatitis (NASH), alcohol associated hepatitis, cholestatic liver disease, hepatocellular carcinoma.
* Clinical hepatic decompensation (i.e., ascites, encephalopathy variceal hemorrhage).
* Solid organ or bone marrow transplantation Note: other protocol defined Inclusion/Exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2025-03-25 (Actual); Primary Completion 2027-06 (Estimated); Study Completion 2028-06 (Estimated)

PRIMARY OUTCOMES:
Percentage of participants with a composite endpoint | Week 24
  Achieving composite endpoint defined as virologic response (undetectable HDV RNA or decline in HDV RNA ≥2 log10 IU/mL) and ALT normalization

SECONDARY OUTCOMES:
Percentage of participants with treatment-emergent adverse events (TEAE) as assessed by DAIDS | Weeks 24, 48, 96, and 120, if applicable
  Frequency and severity of TEAEs and serious AEs
Percentage of participants that achieve that achieve virologic response and ALT normalization | Weeks 24, 48, 96, and 120, if applicable
  Change from baseline in HDV RNA and ALT normalization
Percentage of participants with a composite endpoint by treatment regimen | Weeks 24, 48, 96, and 120, if applicable
  Compare the composite endpoint response (change from baseline HDV RNA and ALT normalization) between weekly versus every 4-week regimen of brelovitug
Percentage of participants with HDV associated liver disease progression | Weeks 24, 48, 96, and 120, if applicable
  Determined by an independent data monitoring committee based on changes in liver stiffness, APRI, CPT/MELD score (cirrhotic), and TEAEs.

CONTACTS AND LOCATIONS:
Overall Officials: Bluejay Therapeutics, Study Director — Bluejay Therapeutics
Locations (38):
- United States (15):
  - 247 Garden Grove, Garden Grove, California
  - 242 Huntington Beach, Huntington Beach, California
  - 252 Long Beach, Long Beach, California
  - 244 Los Angeles, Los Angeles, California
  - 250 Miami, Miami, Florida
  - 251, Illinois, Chicago, Illinois
  - 248 Lowa, Cities in Iowa, Iowa
  - 254 Baltimore, Baltimore, Maryland
  - 241, Massachusetts, Boston, Massachusetts
  - 245 New York, New York, New York
  - 256 New York, New York, New York
  - 253 New York, New York, New York
  - 255 New York, New York, New York
  - 257 Philadelphia, Philadelphia, Pennsylvania
  - 249 San Antonio, San Antonio, Texas
- Australia (3):
  - 102 Melbourne, Melbourne, Victoria
  - 101 Camperdown, Camperdown
  - 104 Liverpool, Liverpool
- Bulgaria (5):
  - 703 Sliven, Sliven, Silven
  - 705 Plovdiv, Plovdiv
  - 702 Bulgaria, Sofia
  - 706 Sofia, Sofia
  - 704 Stara Zagora, Stara Zagora
- Canada (4):
  - 233 Calgary, Calgary, Calgary
  - 234 Alberta, Edmonton, Edmonton
  - 231 Toronto, Toronto, Ontario
  - 235 Montreal, Montreal, Quebec
- Georgia (3):
  - 181 Tbilisi, Tbilisi
  - 183 Tbilisi, Tbilisi
  - 182 Tbilisi, Tbilisi
- Israel (2):
  - 212 Haifa, Haifa, Haifa District
  - 211 Israel, Beersheba
- 901 Chisinau, Chisinau, Moldova
- 001 Auckland, Auckland, New Zealand
- 221 Karachi City, Karachi, Karachi, Pakistan
- 291 Belgrade, Belgrade, Belgrade, Serbia
- 191 Istanbul, Istanbul, Istanbul, Turkey (Türkiye)
- 110 Kyiv, Kyiv, Ukraine

IPD SHARING:
Plan to Share IPD: No